CLINICAL TRIAL: NCT01259843
Title: French National Observatory of Aortic Syndromes
Acronym: ONSAA
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Elbaz Meyer, Assistant Professor, French Cardiology Society
Other Study IDs: 07387
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Acute Aortic Syndrome
Keywords: Acute aortic syndrome
MeSH Terms: conditions — Acute Aortic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Aortic Syndrome: Patients admitted to cardiology, radiology or surgery for a clinical picture suggestive of acute aortic syndrome whose diagnosis was subsequently confirmed in due course of hospitalization by further investigations.

SUMMARY:
The study examined the clinical characteristics and conditions of care for patients with acute aortic syndrome (AAS) that will identify patients at risk for increased morbidity and mortality and provide a basis for the eventual achievement of specific studies on the optimal therapeutic management according to different risk profiles. The aim of the Observatory is to provide a photograph "size" of practices in France at present, both in the larger centers than in smaller and optimize diagnostic and therapeutic currently available by the activation pathways of rational management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age (e) over 18 years old
* Patients with a AAS duly authenticated by further tests
* Patients who consented to participate in the study

Exclusion Criteria:

* Refusal of consent for study participation and ancillary studies
* AAS occurring in the aftermath of a traumatic thoracic
* Diagnosis AAS aside in favor of an alternative diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to cardiology, radiology or surgery for a clinical picture suggestive of acute aortic syndrome whose diagnosis was subsequently confirmed in due course of hospitalization by further investigations.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Etiology of AAS | 1 day
  Measure the respective contribution of each of the etiologies of AAS (aortic dissection type A aortic dissection type B aortic wall hematoma, penetrating atherosclerotic ulcer, aneurysm of the thoracic aorta complicated).

SECONDARY OUTCOMES:
Clinical picture | 1 day
  Identify and define the specific clinical picture of each of these new entities recently dismembered as part of AAS. Indeed, if the clinical presentation of classic aortic dissection A and B is well known, that of other entities, individualized recently, remains poorly described.
Diagnostic tests | 1 day
  Evaluate the performance and the respective roles of the various diagnostic tests including recent acquisitions little or no invasive; Trans thoracic ultrasound, ultrasound and trans esophageal chest scan.

CONTACTS AND LOCATIONS:
Overall Officials: Elbaz Meyer, Principal Investigator — Assistance Publique - Hôpitaux de Paris